CLINICAL TRIAL: NCT01078987
Title: Use of Plasmapheresis for Nephrogenic Fibrosing Dermopathy (NFD)/Nephrogenic Systemic Fibrosis (NSF) and Understanding Its Etiology
Brief Title: Plasmapheresis for Nephrogenic Fibrosing Dermopathy (NFD)/Nephrogenic Systemic Fibrosis (NSF)
Acronym: NFD
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Insufficient recruitment
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 51018
Record Dates: First submitted 2010-02-05; First posted 2010-03-02 (Estimated); Last update posted 2014-11-21 (Estimated); Status verified 2014-11

CONDITIONS: Nephrogenic Fibrosing Dermopathy; Nephrogenic Systemic Fibrosis
Keywords: Nephrogenic Fibrosing Dermopathy (NFD); Nephrogenic Systemic Fibrosis (NSF)
MeSH Terms: conditions — Nephrogenic Fibrosing Dermopathy | interventions — Plasmapheresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1 (Active Comparator): One to three 5-day course of plasma exchange (plasmapheresis)
  Interventions: Procedure: Plasmapheresis
- Group 2 (Active Comparator): One to three 5-day course of plasma exchange (plasmapheresis)
  Interventions: Procedure: Plasmapheresis
- Group 3 (No Intervention): No intervention taken
- Group 4 (Active Comparator): One to three 5-day course of plasma exchange (plasmapheresis)
  Interventions: Procedure: Plasmapheresis

INTERVENTIONS:
Procedure: Plasmapheresis — A course of 5 daily treatments of plasma exchange (plasmapheresis) for one to three courses
  Arms: Group 1; Group 2; Group 4

SUMMARY:
The purpose of this study is to evaluate the pathophysiology of nephrogenic fibrosing dermopathy (NFD)/nephrogenic systemic fibrosis (NSF).

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with NFD/NSF following a kidney transplant
* diagnosed with NFD/NSF following a liver transplant
* NFD/NSF and who have not had a kidney or liver transplant
* diagnosed with NFD/NSF and who have not had a kidney or liver transplant

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2002-02; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Improve elasticity of skin, including increased range of motion of compromised joints due to leathery skin | Assessed two weeks after each monthly course of plasmapheresis

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Baron, MD, Principal Investigator — Loma Linda University Medical Center
Locations (1):
- Loma Linda University Medical Center, Loma Linda, California, United States